CLINICAL TRIAL: NCT06085612
Title: Impact of Significant Carotid Stenosis on Retinal Perfusion Measured Via Automated Retinal Oximetry
Status: Recruiting | Type: Observational
Sponsor: University Hospital Olomouc (Other)
Responsible Party: Principal Investigator, Michal Kral, Principal Investigator, University Hospital Olomouc
Other Study IDs: NW24-06-00380
Record Dates: First submitted 2023-10-09; First posted 2023-10-17 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Stroke, Ischemic; Stenosis, Carotid
Keywords: automated retinal oximetry
MeSH Terms: conditions — Ischemic Stroke; Carotid Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Internal Carotid Artery Stenosis: Group of patients with internal carotid stenosis detected via ultrasound examination.
  Interventions: Diagnostic Test: Automated retinal oximetry
- Non stenotic Internal Carotid Artery: Group of patients without internal carotid stenosis on ultrasound examination.
  Interventions: Diagnostic Test: Automated retinal oximetry

INTERVENTIONS:
Diagnostic Test: Automated retinal oximetry — Non invasive standard examination on automated retinal oximetry.

SUMMARY:
Background: Large vessel carotid stenosis represent significant cause of ischaemic stroke. Indication for surgical revascularisation treatment relies on severity stenosis and clinical symptoms. Mild clinical symptoms such as transient ischemic attack, amaurosis fugax or minor stroke preceded large strokes in only 15% of cases.

Aim: The aim of this prospective study is to evaluate whether retinal perfusion is impacted in significant carotid stenosis. Automated retinal oximetry could be used to better evaluate perfusion in post-stenotic basin. The investigators presume the more stenotic blood vessel, the more reduced retinal perfusion is resulting in adaptive changes such as higher arteriovenous saturation difference due to greater oxygen extraction. This could help broaden the indication spectrum for revascularisation treatment for carotid stenosis.

Methods: The investigators plan to enroll 50 patients a year with significant carotid stenosis and cross-examine them with retinal oximetry. Study group will provide both stenotic vessels and non-stenotic vessels forming the control group. Patients with significant carotid stenosis will undergo an MRI examination to determine the presence of asymptomatic recent ischaemic lesions in the stenotic basin, and the correlation to oximetry parameters.

Statistics: Correlation between the severity of stenosis and retinal oximetry parameters will be compared to the control group of non-stenotic sides with threshold of 70%, respectively 80% and 90% stenosis. Data will be statistically evaluated at the 5% level of statistical significance. Results will be then reevaluated with emphasis on MRI findings in the carotid basin.

Conclusion: This prospective case control study protocol wil be used to launch a trial assessing the relationship between significant carotid stenosis and retinal perfusion measured via automated retinal oximetry.

ELIGIBILITY:
Inclusion Criteria:

Study population will include patients examined in ultrasound laboratory in Neurology department of University Hospital Olomouc, regardless of incidental finding of stenosis, examination due to acute symptoms or regular checkup of known stenosis.

Exclusion Criteria:

* patients unable undergo ophthalmological examination properly, especially on automated retinal oximetry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will include patients examined in Neurosonological laboratory in Neurology department of University Hospital Olomouc,
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Arterio-venous oxygen difference in retinal blood vessels measured by automated retinal oximetry. | 2028
  To establish whether arterio-venous difference in the stenotic basin increases with the severity of stenosis and/or these changes vary depending on the severity of stenosis.

SECONDARY OUTCOMES:
Correlation with MRI ischaemic lesions | 2029
  with clinically symptomatic and asymptomatic carotid stenosis correlated to MRI findings of ipsilateral ischaemic lesions in the stenotic basin.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Olomouc, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Polidar P, Paskova B, Karhanova M, Sin M, Dornak T, Schreiberova Z, Divisova P, Veverka T, Franc D, Sanak D, Kral M. Study protocol - Prospective case-control trial - Impact of significant carotid stenosis on retinal perfusion measured with automated retinal oximetry. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2025 Mar;169(1):66-71. doi: 10.5507/bp.2023.052. Epub 2024 Jan 3. PMID 38192247